CLINICAL TRIAL: NCT05395572
Title: The Effects of Kinesio® Tape on Neck Pain and Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Dakota State University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: IRB0003476
Record Dates: First submitted 2021-06-02; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2021-06

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tape (Experimental): Kinesio tape will be applied to the neck to help facilitate underactive muscles and ROM will be assessed
  Interventions: Device: Kinesio® Tape
- Control (No Intervention): ROM will be assessed before tape application to determine any changes

INTERVENTIONS:
Device: Kinesio® Tape — In order to increase the activity of underactive muscles, the tape is applied from origin to insertion with a 15-25% tension. The Kinesio® Tape mechanical muscle correction will be performed with one Y-strip of Kinesio® Tape over the bilateral cervical multifidus and semispinalis cervicis muscles, while also including portions of other cervical extensor muscles (the semispinalis capitis, splenius cervicis, levator scapulae, upper trapezius, longus coli, and splenius capitis).
  Arms: Tape

SUMMARY:
This study is a within-subjects design; therefore, the participant will serve as their own control. Participants will be included in the study if they have neck pain or disability defined by a score of more than 14 on the Neck Disability Index. They will be excluded if they have any diagnosed disc pathology. A mask-associated pain questionnaire will be completed by the participants prior to the study to determine their perceived effect of mask-wearing on neck pain. This questionnaire is adapted from the HAPPE study on mask-associated headache pain. A baseline pain rating will be recorded a numerical pain scale. Next, active cervical range of motion will be measured, three times in each direction to be averaged. A pain rating will be recorded for pain during cervical motion. Kinesio® Tape will be applied to activate the cervical extensor muscles. The participant will sit with the tape on for 20 minutes, then active cervical range of motion and pain will be recored again.

ELIGIBILITY:
Inclusion Criteria:

* Neck Disability Index Score of more than 14

Exclusion Criteria:

* cervical disc pathology or injury
* previous neck surgery
* prior history of general medical conditions involving joints, muscles, bones or connective tissue such as fibromyalgia, osteoporosis, etc.
* an NDI score of less than 14 or more than 24
* reported allergies to Kinesio® Tex Tape or any other adhesive material
* any contraindications for the usage of Kinesio® Tape

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-17 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index | 1 day
  Patient-reported neck pain
Headaches Associated With Personal Protective Equipment | 1 day
  Mask associated pain questionnaire
Dartfish | 20 minutes
  2-dimensional motion analysis

CONTACTS AND LOCATIONS:
Locations (1):
- North Dakota State University, Fargo, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No